CLINICAL TRIAL: NCT02555410
Title: A Pivotal, Phase II Trial of Detecting Generalized Tonic-Clonic Seizures With a Seizure Detection and Warning System in Epilepsy Patients
Brief Title: Seizure Detection and Warning System in Epilepsy Patients
Status: Completed | Type: Observational
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Other Study IDs: 3.01P
Record Dates: First submitted 2015-02-13; First posted 2015-09-21 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy; Generalized Tonic-Clonic Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Sentinel Seizure Detection and Warning System: To test the usability of the Brain Sentinel Seizure Detection and Warning System(also known as the SPEAC system) in a patient home setting.
  Interventions: Device: Brain Sentinel Seizure Detection and Warning System

INTERVENTIONS:
Device: Brain Sentinel Seizure Detection and Warning System — A sEMG based automated seizure detection and warning system worn on the biceps
  Other Names: SPEAC System

SUMMARY:
This is a phase III, pilot, prospective study of an Electromyography (EMG) based seizure detection system for detecting Generalized Tonic-Clonic Seizures (GTCS) in the home.

DETAILED DESCRIPTION:
The Brain Sentinel™ Seizure Detection and Warning System is intended for monitoring children and adults with a history or significant risk of generalized tonic-clonic seizures in the home or healthcare facilities, during the titration or withdrawal of anti-epileptic drugs, and for continuous monitoring (night time or any other time of day) of individuals due to their history or risk of generalized tonic-clonic seizures. The device will withstand activities of daily living including showers and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization.
2. Male or female between the ages of 2-99.
3. Has an upper arm circumference which is adequate for proper fit of the EMG monitor (at least 14cm).
4. Be able to tolerate wearing the device on the upper arm.
5. If female and of childbearing potential, has a negative pregnancy test.
6. Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
7. Subject and/or Primary Caregiver must be competent to follow all study procedures.
8. Is able to read, speak and understand English.

Exclusion Criteria:

1. Does not have a documented history of generalized seizures.
2. The subject's upper arm circumference not adequate for proper fit of the EMG monitor (less than 14cm)
3. Pregnant female
4. Subject/Caregiver is unable to provide consent.
5. Subject/Caregiver is not competent to follow home study procedures.
6. The subject is homeless or in a home without a power supply.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Test the function of the system including ability to acquire EMG signal, analyze and successfully transmit the analysis to the base station, and identify and transmit all alert conditions. | up to 1 month
  The overall usability and technical features will be assessed through questionnaires and surveys as the Seizure Detection and Warning System will be used within a home setting.

SECONDARY OUTCOMES:
Compare the accuracy of the EMG based system's log to the subject's seizure diary | up to one month
  Comparison of the subject's seizure diary to the EMG based seizure detection system's seizure logs will help determine overall function.

CONTACTS AND LOCATIONS:
Overall Officials: Jose E. Cavazos, MD, PhD, Principal Investigator — Brain Sentinel
Locations (1):
- Jose' E. Cavazos, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No